CLINICAL TRIAL: NCT05932641
Title: A Phase I Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD3152 in Healthy Japanese Adults
Brief Title: Study of AZD3152 Intramuscular Injection or Intravenous Infusion in Healthy Japanese Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D7000C00007
Record Dates: First submitted 2023-05-15; First posted 2023-07-06 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: COVID-19, SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This is a Phase I, randomised, double-blind, placebo controlled study evaluating the safety, tolerability, PK and PD of AZD3152 in healthy Japanese adult participants, 18 to 55 years of age. Approximately 24 healthy participants will be randomised at up to 2 study sites in a ratio of 6:2 in each cohort to either AZD3152 or placebo administered IM or IV, across 3 fixed-dose cohorts. To participants who will receive the IMP via IM injection (Cohorts 1 and 2), the IMP will be given as a direct anterolateral thigh IM administration of AZD3152 or placebo. To participants who will receive the IMP via IV infusion (Cohort 3), the IMP will be administered as an IV infusion containing AZD3152 or placebo. The randomisation of Cohort 2 and 3 should be performed sequentially.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Cohort 1 - AZD3152 300 mg IM direct anterolateral thigh injection (Experimental)
  Interventions: Biological: AZD3152 (Cohort 1)
- Cohort 1 - Placebo IM direct anterolateral thigh injection (Placebo Comparator)
  Interventions: Biological: Placebo (Cohort 1)
- Cohort 2 - AZD3152 600 mg IM direct anterolateral thigh injection (Experimental)
  Interventions: Biological: AZD3152 (Cohort 2)
- Cohort 2 - Placebo direct anterolateral thigh injection (Placebo Comparator)
  Interventions: Biological: Placebo (Cohort 2)
- Cohort 3 - AZD3152 1200 mg IV administration (Experimental)
  Interventions: Biological: AZD3152 (Cohort 3)
- Cohort 3 - Placebo IV administration (Placebo Comparator)
  Interventions: Biological: Placebo (Cohort 3)

INTERVENTIONS:
Biological: AZD3152 (Cohort 1) — Single dose of AZD3152 300 mg IM on Visit 2 Day 1
  Arms: Cohort 1 - AZD3152 300 mg IM direct anterolateral thigh injection
Biological: Placebo (Cohort 1) — Single dose of Placebo IM on Visit 2 Day 1
  Arms: Cohort 1 - Placebo IM direct anterolateral thigh injection
Biological: AZD3152 (Cohort 2) — Single dose of AZD3152 600 mg IM on Visit 2 Day 1
  Arms: Cohort 2 - AZD3152 600 mg IM direct anterolateral thigh injection
Biological: Placebo (Cohort 2) — Single dose of Placebo IM on Visit 2 Day 1
  Arms: Cohort 2 - Placebo direct anterolateral thigh injection
Biological: AZD3152 (Cohort 3) — Single dose of AZD3152 1200 mg IV on Visit 2 Day 1
  Arms: Cohort 3 - AZD3152 1200 mg IV administration
Biological: Placebo (Cohort 3) — Single dose of Placebo IM on Visit 2 Day 1
  Arms: Cohort 3 - Placebo IV administration

SUMMARY:
AZD3152 is being evaluated for administration to prevent COVID-19. This Phase I study will gather important information on the safety and tolerability of AZD3152 as well as relevant data on the PK, PD (as the neutralising responses against SARS-CoV-2) profile and the generation of ADA to AZD3152.

DETAILED DESCRIPTION:
This is a Phase I, randomised, double-blind, placebo controlled study evaluating the safety, tolerability, PK and PD of AZD3152 in healthy Japanese adult participants, 18 to 55 years of age. Approximately 24 healthy participants will be randomised at up to 2 study sites.

ELIGIBILITY:
Inclusion Criteria:

* Japanese men and women and 18 to 55 years of age inclusive, at the time of signing the informed consent.
* No positive results of SARS-CoV-2 NAT and/or rapid antigen tests.
* Healthy participants by medical history, physical examination, baseline safety laboratory studies, and screening parameters, according to the judgement of the investigators, with no concomitant disease or concomitant medication.
* ECG without clinically significant abnormalities.
* Able to complete the Follow-up Period through Day 361 as required by the protocol.
* Body weight ≥ 45 kg and ≤ 110 kg and BMI ≥ 18.0 to ≤ 30.0 kg/m2.

Exclusion Criteria:

* Known hypersensitivity to any component of the IMP.
* History of allergic disease or reactions likely to be exacerbated by any component of the IMP.
* Previous hypersensitivity, infusion related reaction or severe adverse reaction following administration of mAbs.
* Fever above 38.0°C on day prior to or on day of randomisation/dosing.
* AST, ALT or serum creatinine above ULN; bilirubin and ALP >1.5 × ULN.
* Any vaccination except for COVID-19 vaccine (e.g., inactivated influenzae vaccine) planned.
* SARS CoV-2 or COVID-19:

Receipt of a COVID-19 vaccine within 3 months. COVID-19 infection within 3 months prior.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of AZD3152 - AEs | Up to Visit 9 (Day 91)
  Occurrence of AEs collected up to Visit 9 (Day 91)
To evaluate the safety and tolerability of AZD3152 - SAEs, MAAEs, and AESIs | Up to Visit 12 (Day 361)
  Occurrence of SAEs, MAAEs, and AESIs collected up to Visit 12 (Day 361)
To evaluate the safety and tolerability of AZD3152 - Blood pressure | Up to Visit 7 (Day 29)
  The following variables will be collected:
  * Systolic Blood pressure
  * Diastolic Blood pressure
To evaluate the safety and tolerability of AZD3152 - Pulse rate | Up to Visit 7 (Day 29)
  Pulse rate will be collected
To evaluate the safety and tolerability of AZD3152 - Axillary temperature | Up to Visit 7 (Day 29)
  Axillary temperature will be collected
To evaluate the safety and tolerability of AZD3152 - Respiratory rate | Up to Visit 7 (Day 29)
  Respiratory rate will be collected
To evaluate the safety and tolerability of AZD3152 - PR Interval, QRS Duration, QT Interval, QTcF Interval and RR Interval | Up to Visit 7 (Day 29)
  PR Interval, QRS Duration, QT Interval, QTcF Interval and RR Interval will be recorded
To evaluate the safety and tolerability of AZD3152 - Heart rate | Up to Visit 7 (Day 29)
  Heart rate will be recorded
To characterise the Serum Pharmacokinetics of AZD3152 - Concentration at the end of infusion (Ceoi) (after intravenous only) | Up to Visit 12 (Day 361)
  AZD3152 concentration over time and Pharmacokinetics parameters
To characterise the Serum Pharmacokinetics of AZD3152 - Maximum concentration (Cmax) | Up to Visit 12 (Day 361)
  AZD3152 concentration over time and Pharmacokinetics parameters
To characterise the Serum Pharmacokinetics of AZD3152 - Time to maximum concentration (tmax) | Up to Visit 12 (Day 361)
  AZD3152 concentration over time and Pharmacokinetics parameters
To characterise the Serum Pharmacokinetics of AZD3152 - Terminal half-life (t½) | Up to Visit 12 (Day 361)
  AZD3152 concentration over time and Pharmacokinetics parameters
To characterise the Serum Pharmacokinetics of AZD3152 - Area under the concentration-time curve at the last measured time point (AUClast) | Up to Visit 12 (Day 361)
  AZD3152 concentration over time and Pharmacokinetics parameters
To characterise the Serum Pharmacokinetics of AZD3152 - Area under the concentration-time curve from time zero extrapolated to infinity (AUCinf) | Up to Visit 12 (Day 361)
  AZD3152 concentration over time and Pharmacokinetics parameters
To evaluate the safety and tolerability of AZD3152 - Haematology - White blood cell count | Up to Visit 7 (Day 29)
  The following will be collected:
  - White blood cell count
To evaluate the safety and tolerability of AZD3152 - Haematology - Red blood cell count | Up to Visit 7 (Day 29)
  The following will be collected:
  - Red blood cell count
To evaluate the safety and tolerability of AZD3152 - Haematology - Haemoglobin | Up to Visit 7 (Day 29)
  The following will be collected:
  - Haemoglobin
To evaluate the safety and tolerability of AZD3152 - Haematology - Haematocrit | Up to Visit 7 (Day 29)
  The following will be collected:
  - Haematocrit
To evaluate the safety and tolerability of AZD3152 - Haematology - Mean corpuscular volume | Up to Visit 7 (Day 29)
  The following will be collected:
  - Mean corpuscular volume
To evaluate the safety and tolerability of AZD3152 - Haematology - Mean corpuscular haemoglobin | Up to Visit 7 (Day 29)
  The following will be collected:
  - Mean corpuscular haemoglobin
To evaluate the safety and tolerability of AZD3152 - Haematology - Mean corpuscular haemoglobin concentration | Up to Visit 7 (Day 29)
  The following will be collected:
  - Mean corpuscular haemoglobin concentration
To evaluate the safety and tolerability of AZD3152 - Haematology - Neutrophils absolute count | Up to Visit 7 (Day 29)
  The following will be collected:
  - Neutrophils absolute count
To evaluate the safety and tolerability of AZD3152 - Haematology - Lymphocytes absolute count | Up to Visit 7 (Day 29)
  The following will be collected:
  - Lymphocytes absolute count
To evaluate the safety and tolerability of AZD3152 - Haematology - Monocytes absolute count | Up to Visit 7 (Day 29)
  The following will be collected:
  - Monocytes absolute count
To evaluate the safety and tolerability of AZD3152 - Haematology - Eosinophils absolute count | Up to Visit 7 (Day 29)
  The following will be collected:
  - Eosinophils absolute count
To evaluate the safety and tolerability of AZD3152 - Haematology - Basophils absolute count | Up to Visit 7 (Day 29)
  The following will be collected:
  - Basophils absolute count
To evaluate the safety and tolerability of AZD3152 - Haematology - Platelets | Up to Visit 7 (Day 29)
  The following will be collected:
  - Platelets
To evaluate the safety and tolerability of AZD3152 - Haematology - Reticulocytes absolute count | Up to Visit 7 (Day 29)
  The following will be collected:
  - Reticulocytes absolute count
To evaluate the safety and tolerability of AZD3152 - Serum Clincal Chemistry - Sodium | Up to Visit 7 (Day 29)
  The following will be collected:
  - Sodium
To evaluate the safety and tolerability of AZD3152 - Serum Clincal Chemistry - Potassium | Up to Visit 7 (Day 29)
  The following will be collected:
  - Potassium
To evaluate the safety and tolerability of AZD3152 - Serum Clincal Chemistry - Blood urea nitrogen | Up to Visit 7 (Day 29)
  The following will be collected:
  - Blood urea nitrogen
To evaluate the safety and tolerability of AZD3152 - Serum Clincal Chemistry - Creatinine and estimated glomerular filtration rate | Up to Visit 7 (Day 29)
  The following will be collected:
  - Creatinine and estimated glomerular filtration rate
To evaluate the safety and tolerability of AZD3152 - Serum Clincal Chemistry - Albumin | Up to Visit 7 (Day 29)
  The following will be collected:
  - Albumin
To evaluate the safety and tolerability of AZD3152 - Serum Clincal Chemistry - Calcium | Up to Visit 7 (Day 29)
  The following will be collected:
  - Calcium
To evaluate the safety and tolerability of AZD3152 - Serum Clincal Chemistry - Phosphate | Up to Visit 7 (Day 29)
  The following will be collected:
  - Phosphate
To evaluate the safety and tolerability of AZD3152 - Serum Clincal Chemistry - Glucose | Up to Visit 7 (Day 29)
  The following will be collected:
  - Glucose
To evaluate the safety and tolerability of AZD3152 - Serum Clincal Chemistry - C reactive protein | Up to Visit 7 (Day 29)
  The following will be collected:
  - C reactive protein
To evaluate the safety and tolerability of AZD3152 - Alkaline phosphatase | Up to Visit 7 (Day 29)
  The following will be collected:
  - Alkaline phosphatase
To evaluate the safety and tolerability of AZD3152 - Serum Clincal Chemistry - Alanine aminotransferase | Up to Visit 7 (Day 29)
  The following will be collected:
  - Alanine aminotransferase
To evaluate the safety and tolerability of AZD3152 - Serum Clincal Chemistry - Aspartate aminotransferase | Up to Visit 7 (Day 29)
  The following will be collected:
  - Aspartate aminotransferase
To evaluate the safety and tolerability of AZD3152 - Serum Clincal Chemistry - Gamma glutamyl transpeptidase | Up to Visit 7 (Day 29)
  The following will be collected:
  - Gamma glutamyl transpeptidase
To evaluate the safety and tolerability of AZD3152 - Serum Clincal Chemistry - Total bilirubin | Up to Visit 7 (Day 29)
  The following will be collected:
  - Total bilirubin
To evaluate the safety and tolerability of AZD3152 - Serum Clincal Chemistry - Unconjugated bilirubin | Up to Visit 7 (Day 29)
  The following will be collected:
  - Unconjugated bilirubin
To evaluate the safety and tolerability of AZD3152 - Serum Clincal Chemistry - Conjugated bilirubin | Up to Visit 7 (Day 29)
  The following will be collected:
  - Conjugated bilirubin
To evaluate the safety and tolerability of AZD3152 - Serum Clincal Chemistry - Creatine kinase | Up to Visit 7 (Day 29)
  The following will be collected:
  - Creatine kinase
To evaluate the safety and tolerability of AZD3152 - Serum Clincal Chemistry - Troponin T and I | Up to Visit 7 (Day 29)
  The following will be collected:
  - Troponin T and I
To evaluate the safety and tolerability of AZD3152 - Urinalysis - Glucose | Up to Visit 7 (Day 29)
  The following will be collected:
  - Glucose
To evaluate the safety and tolerability of AZD3152 - Urinalysis - Blood | Up to Visit 7 (Day 29)
  The following will be collected:
  - Blood
To evaluate the safety and tolerability of AZD3152 - Urinalysis - Microscopy | Up to Visit 7 (Day 29)
  The following will be collected:
  - Microscopy
To evaluate the safety and tolerability of AZD3152 - Urinalysis - Protein | Up to Visit 7 (Day 29)
  The following will be collected:
  - Protein
To evaluate the safety and tolerability of AZD3152 - Coagulation - International normalised ratio | Up to Visit 7 (Day 29)
  The following will be collected:
  - International normalised ratio
To evaluate the safety and tolerability of AZD3152 - Coagulation - Activated partial thrombin time | Up to Visit 7 (Day 29)
  The following will be collected:
  - Activated partial thrombin time
To evaluate the safety and tolerability of AZD3152 - Coagulation - Prothrombin time | Up to Visit 7 (Day 29)
  The following will be collected:
  - Prothrombin time

SECONDARY OUTCOMES:
To evaluate the Anti-Drug Antibody responses to AZD3152 in serum | Up to Visit 12 (Day 361)
  Incidence of Anti-Drug Antibody to AZD3152 in serum
The serum neutralising responses against SARS-CoV-2 using geometric mean titer (GMT) and geometric mean fold rise (GMFR) from baseline | Up to Visit 12 (Day 361)
  Blood samples as neutralising responses against SARS-CoV-2 in serum will be collected

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home